CLINICAL TRIAL: NCT06888128
Title: The STARLIGHT Protocol: State-Funded Trial Assessing Recovery and Long-Term Impact of Guided Psilocybin for Healing Trauma
Brief Title: State-Funded Trial Assessing Recovery and Long-Term Impact of Guided Psilocybin for Healing Trauma
Acronym: STARLIGHT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Texas Department of State Health Services (Other); Usona Institute (Other); AIM Youth Mental Health (Unknown)
Responsible Party: Principal Investigator, Lynnette Astrid Averill, Associate Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-50300
Record Dates: First submitted 2025-02-21; First posted 2025-03-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: PTSD
Keywords: PTSD; veterans; psilocybin; trauma; psychedelic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Psilocybin-assisted therapy (Experimental): Participants will enter a 5-week participation phase, which includes 3 preparatory sessions, 2 dosing days, and 4 integration sessions.
  Interventions: Drug: Psilocybin 15mg; Drug: Psilocybin 25mg

INTERVENTIONS:
Drug: Psilocybin 15mg — Each participant will have a low dose (15 mg) psilocybin session to establish basic skills with session format, psilocybin effects, and continue to build rapport with session facilitators. Given the potential intensity of the psilocybin and the reality of experiencing significant trauma memories, the purpose of the first psilocybin session is to familiarize participants with the drug effects that may be encountered at a higher dose of psilocybin. The first psilocybin session will also allow for assessment of both the suitability of each participant to the study procedures and drug effects, and the safety of administering a higher dose to each participant.
Drug: Psilocybin 25mg — The second psilocybin session will utilize a high dose (25mg) and take place approximately 2 weeks after the first psilocybin session.

SUMMARY:
The principal investigator for this study plans to build upon the psilocybin-assisted therapy intervention used in prior completed trials to conduct an open-label trial of two psilocybin administration sessions combined with psychotherapy to investigate the safety, tolerability, and clinical efficacy of psilocybin-assisted therapy for the treatment of PTSD in US Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Be a United States Military Veteran
* Have at least a high-school level of education or equivalent (e.g. GED).
* Have a current DSM-5 diagnosis of Post-traumatic Stress Disorder
* Have a CAPS-5 total severity score of ≥23 at baseline
* SSRIs will be allowable so long as participants are on a stable regimen for a period of 3 months.
* Concurrent psychotherapy is allowed if the type and frequency of the therapy has been stable for at least 2 months prior to screening and is expected to remain stable during participation in the study.
* Be medically stable as determined by screening for medical problems via a personal interview, a medical questionnaire, a physical examination, an electrocardiogram (ECG), and routine medical blood and urinalysis laboratory tests
* No use of hallucinogens in the past 3 months and no history of regular or frequent use of hallucinogens

Exclusion Criteria:

* General medical exclusion criteria:

  * Individuals who are pregnant or nursing; individuals who are of child-bearing potential and sexually active who are not practicing a highly effective means of birth control
  * Individuals with partners of childbearing potential who are sexually active and not practicing a highly effective means of contraception
  * Cardiovascular conditions: coronary artery disease, stroke, angina, uncontrolled hypertension, a clinically significant ECG abnormality (e.g., atrial fibrilation), prolonged QTc interval (i.e., QTc > 450 msec), artificial heart valve, or TIA in the past year • Systolic blood pressure (SBP) > 139 mm HG; diastolic blood pressure (DBP) > 89 mm HG; heart rate (HR) > 90 bpm.
  * Epilepsy with history of seizures
  * Insulin-dependent diabetes; if taking oral hypoglycemic agent, then no history of symptoms of hypoglycemia
* Psychiatric Exclusion Criteria:

  * Current or past history of meeting DSM-5 criteria for schizophrenia spectrum or other psychotic disorders (except substance/medication-induced or due to another medical condition), or Bipolar I or II Disorder
  * Current or history within six months of meeting DSM-5 criteria for a moderate or severe alcohol, tobacco, caffeine, or other drug use disorder; if a regular smoker, they must agree to use a nicotine patch on the day of dosing as smoking will not be allowed on these sessions
  * Have a first degree relative with schizophrenia spectrum or other psychotic disorders including substance/medication-induced or due to another medical condition
  * Risk for acute suicidality as determined by clinician judgment (C-SSRS)
  * Has a psychiatric condition which precludes the establishment of therapeutic rapport as evidenced by long-term patterns of unstable relationships, history of significant stress-related paranoia, and identity disturbances
  * History of a medically significant suicide attempt
  * Current MAOI antidepressant use

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Safety of psilocybin-assisted therapy for PTSD | Baseline to 6-month follow up
  Safety as measured by Adverse Event Reporting
Safety of psilocybin-assisted therapy for PTSD | Baseline to 6-month follow up
  Safety as measured by changes in suicidal ideation on the Columbia Suicide Safety Rating Scale (CSSRS). This section of the measure is assessed on a scale of 0 to 25, with higher scores indicating greater intensity of suicidal ideation.
Efficacy of psilocybin-assisted therapy for PTSD | Baseline to 6-month follow up
  Change in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) score. This measure is assessed on a scale of 0 to 80, with higher scores reflecting increased severity of PTSD symptoms.

SECONDARY OUTCOMES:
Self-reported clinical efficacy of psilocybin-assisted therapy for PTSD symptoms | Baseline to 6-month follow up
  Change in self-reported PTSD Checklist 5 (PCL-5) scores. This measure is assessed on a scale of 0 to 80, with higher scores reflecting increased severity of PTSD symptoms.
Self-reported clinical efficacy of psilocybin-assisted therapy for depressive symptoms | Baseline to 6-month follow up
  Changes in self-reported Quick Inventory of Depression Severity (QIDS) scores. This measure is assessed on a scale of 0 to 27, with higher scores reflecting increased severity of depressive symptoms.
Self-reported clinical efficacy of psilocybin-assisted therapy for anxiety symptoms | Baseline to 6-month follow up
  Changes in self-reported Generalized Anxiety Disorder-7 (GAD-7) scores. This measure is assessed on a scale of 0 to 21, with higher scores reflecting increased severity of anxiety symptoms.

OTHER OUTCOMES:
Changes in Resting-State Functional Connectivity | Baseline to 6-month follow up
  The effect of psilocybin-assisted therapy on functional connectivity networks using resting-state functional magnetic resonance imaging (MRI)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-11): https://cdn.clinicaltrials.gov/large-docs/28/NCT06888128/Prot_SAP_000.pdf
  • Informed Consent Form (2024-12-11): https://cdn.clinicaltrials.gov/large-docs/28/NCT06888128/ICF_001.pdf